CLINICAL TRIAL: NCT06899763
Title: Single-Cell Profiling of Liver-infiltrating Immune Cells of Patients with NASH- and Virus-related HCC: Implications for Immunotherapy
Acronym: 1003rcr2022_72
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefania Mantovani, Researcher, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 1003rcr2022_72
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC); MASLD-HCC; HCV_HCC
Keywords: hepatocellular carcinoma; MASLD; HCV
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with MASLD-related HCC: The cohort is composed of patients with MASLD-related HCC. MASLD, previously termed non-alcoholic fatty liver disease (NAFLD), is defined as steatotic liver disease (SLD) in the presence of one or more cardiometabolic risk factor(s) and the absence of harmful alcohol intake (Rinella ME, Lazarus JV, Ratziu V, et al. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. J Hepatol. 2023;79(6):1542-1556. doi:10.1016/j.jhep.2023.06.003).
- patients with HCV-related HCC: The cohort is composed of patients with HCV-related HCC.

SUMMARY:
The goal of this observational study is to learn about the the immune landscape of HCC arising from different etiology, such as MASLD and viral hepatitis, at single cell level. The main question it aims to answer is:

Which are the immune signatures and pathways linked to MASLD- or virus-related HCC and what could be the best targets for immunotherapy?

DETAILED DESCRIPTION:
The TME is infiltrated by several populations of immune cells, among which effector cytotoxic T and NK cells mediate tumor immuno-surveillance. By contrast, inhibitory subpopulations, including CD4+ regulatory T cells and tumor-associated myeloid cells and macrophages, can counteract immune responses and favor tumor growth. Some studies have recently deciphered the composition of the TME in HCC regardless of etiology.

In order to unveil differences in the infiltrating immune cells associated with MASL- and virus-related HCC we propose the following:

1. Patient enrollment, sample collection, processing and biobanking.
2. Analysis of non-tumoral liver- and tumor-infiltrating immune cells of MASLD- and virus-related HCC by scRNA-seq.
3. Intervention on newly discovered etiology-associated immune mechanisms identified in the present study to unlock/boost anti-tumor cytotoxic NK and T cell functions.

One major asset to this study is the availability of cryopreserved surgical specimens obtained from previously collected liver resections for HCC, consisting of patients with chronic HBV and HCV infections, as well as MASLD. Infiltrating mononuclear cells are cryopreserved live in 90% fetal calf serum/DMSO. This will provide an immediate availability of biological material from well characterized patients and will serve as a training set that shall be validated in a subsequent prospective cohort that will be recruited during the entire study. To this end, internal and external collaborating surgical units plan to collect approximately 20 virus-related HCC patients with chronic hepatitis B- or C virus infection and 20 MASLD-related HCC untreated at the time of the study. Complete clinical data will be collected in a dedicated database. Peripheral blood mononuclear cells (PBMC) will be obtained by Ficoll-Paque gradient and cryopreserved. Serum will be separated from whole blood and preserved at -80°C. PBMC and serum derived from patients will be collected for biobanking. Surgically resected tumor specimens and matched non adjacent non-tumoral tissue will be mechanically and enzymatically dissociated with the human Tumor Dissociation Kit by gentleMACS Dissociator to separate liver- and tumor-infiltrating mononuclear cells (LIM and TIM respectively). Short-term 2D culture will be established from each patient's tumor tissue.

To investigate which cellular subsets and pathways are associated with MASLD- or virus-related HCC we will take advantage of scRNA-seq technology that provides a detailed view on differences in gene expression between cell types or transcriptome heterogeneity across cells of the same type. We will perform scRNA-seq of CD45+ LIM and TIM. To this end, we will isolate CD45+ cells from LIM and TIM by flow cytometry cell sorting. To prepare libraries from single cells we will use the micro-well based BD Rhapsody platform. Next, sequencing of the whole transcriptome will be performed on an Illumina sequencing platform. We are planning to perform sequencing from 4 to 6 patients for MASLD- and virus-related HCC. The SeqGeq™ desktop bioinformatics platform will be used to analyze scRNA-seq data to detect highly variable genes, perform PCA, graph-based clustering, and t-SNE. The goal will be to compare the transcriptional profiles of LIM and TIM derived from HCC with different etiology, as well as comparing LIM and TIM of the same patient. Differential gene expression analysis will be conducted with a log-scaled fold change ≥1.5 and P value <0.05. Comparison of gene signature expression between two groups of cells will be performed using unpaired two-tailed Wilcoxon rank-sum tests. Since single-cell transcriptomics generally provides a massive amount of information, special attention will initially be paid to genes involved in the metabolic status, associated with cytotoxic responses and release of cytotoxic granules, encoding for activating and inhibitory receptors and for immunosuppressive/activatory molecules.

This approach should lead to the definition of which cellular subsets of LIM and TIM and which pathways define the TME of MASLD- and virus-related HCC. Special attention will be paid on cellular subset deputized to immune surveillance, such as NK and T cells and on ligand-activating receptor axes involved in tumor recognition.

Once a panel of key etiology-associated immune mechanisms will be identified, it will be important i) to validate findings in a larger cohort and ii) to target the most promising newly discovered pathways to restore anti-tumor cytotoxic NK and T cell functions.

i) Data will be validated on a higher number of patients, i.e. measuring gene expression by real-time PCR and analyzing immune infiltrate by flow cytometry. ii) We will perform in vitro experiments in which LIM and TIM will be co-cultured with autologous primary HCC cells in the presence of molecules and/or mAbs that interfere on selected pathways. A combination of experimental data, bioinformatic analysis and an extensive revision of the literature will be crucial to identify the best druggable spot to be used for our purpose. For instance, mAbs will be used to intercept immunosuppressive molecules and abrogate their effect, or to stimulate activating pathways, or, alternatively, to block inhibitory receptors. Gene expression analysis as well as flow cytometry, measuring the cytotoxic granules and cytokines released from cytotoxic cells, will be employed to assess NK and T cell function.

ELIGIBILITY:
Inclusion criteria:

* HCV-related HCC or MASLD-related HCC
* age: ≥ 18 years, ≤ 90 years
* Signature of the informed consent

Esclusion criteria:

* Concomitant pathologies with a life expectancy of less than 12 months
* Autoimmune or chronic inflammatory diseases
* Treatment with atezolizumab, bevacizumab, sorafenib, lenvatinib, regorafenib, cabozantinib, checkpoint inhibitors, tyrosine kinase inhibitors, or anti-VEGF therapies
* Other ongoing extrahepatic malignancies or those diagnosed within the last 3 years, except for tumors resected with curative intent and with no evidence of disease recurrence for >3 years prior to the signing of informed consent, and considered at low risk of recurrence
* HIV infection
* Lack of patient cooperation and failure to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of MASLD-related HCC or HCV-related HCC
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of differentially expressed genes (DEGs) among different patients in the various cellular clusters identified, using scRNA-seq. | until the end of the study, approximatively 2 years
  scRNA-seq will provide data to perform cell type annotation. For each cluster DEG will be identify through bioinformatic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No